CLINICAL TRIAL: NCT02096744
Title: A Randomized, Double-blind Study Designed to Assess the Bioequivalence and Adhesion Properties of Transdermal Clonidine-VistanexTM Compared to Transdermal Clonidine-Oppanol® Following Transdermal Administration in Healthy Male and Female Volunteers
Brief Title: Bioequivalence of Two Transdermal Clonidine Administrations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 253.2486
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — Clonidine

ARMS (3):
- Catapres-TTS-3 crossover 1 (Experimental): subject to receive 0.3 mg/24 hr Catapres-TTS-3 Oppanol (T1) first, followed by Catapres-TTS-3 Vistanex (R1)
  Interventions: Drug: Intervention 1: Catapres-TTS-3; Drug: Intervention 2: Catapres-TTS-3
- Catapres-TTS-3 crossover 2 (Experimental): subject to receive 0.3 mg/24 hr Catapres-TTS-3 Vistanex (R1) first, followed by Catapres-TTS-3 Oppanol (T1)
  Interventions: Drug: Intervention 1: Catapres-TTS-3; Drug: Intervention 2: Catapres-TTS-3
- Catapres-TTS-1 crossover 1 (Experimental): subject to receive 0.1 mg/24 hr Catapres-TTS-1 with Oppanol (T2) and Vistanex (R2) simultaneously
  Interventions: Drug: Catapres-TTS-1

INTERVENTIONS:
Drug: Catapres-TTS-1 — Catapres-TTS-1 Oppanol
  Arms: Catapres-TTS-1 crossover 1
Drug: Intervention 1: Catapres-TTS-3 — Catapres-TTS-3 Oppanol
  Arms: Catapres-TTS-3 crossover 1
Drug: Intervention 1: Catapres-TTS-3 — Catapres-TTS-3 Oppanol
  Arms: Catapres-TTS-3 crossover 2
Drug: Intervention 2: Catapres-TTS-3 — Catapres-TTS-3 Vistanex
  Arms: Catapres-TTS-3 crossover 2
Drug: Catapres-TTS-1 — Catapres-TTS-1 Vistanex
  Arms: Catapres-TTS-1 crossover 1
Drug: Intervention 2: Catapres-TTS-3 — Catapres-TTS-3 Vistanex
  Arms: Catapres-TTS-3 crossover 1

SUMMARY:
To establish the bioequivalence and adhesion properties of transdermal clonidine prepared with Oppanol® brands of polyisobutylene (PIB) vs. transdermal clonidine prepared with VistanexTM brands of polyisobutylene (PIB) in healthy male and female volunteers.

ELIGIBILITY:
Inclusion criteria:

1. A complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age greater than or equal to 18 and Age less than or equal to 65 years
3. BMI greater than or equal to 18.5 and BMI less than or equal to 32.0 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study
5. Male subjects, or females who meet any of the following criteria from at least 30 days before the first study drug administration and until 30 days after trial completion:

   * Using adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral contraceptives, intrauterine device (IUD)
   * Sexually abstinent
   * Have a vasectomised sexual partner (vasectomy at least one year prior to enrolment)
   * Surgically sterilised (including hysterectomy)
   * Postmenopausal defined as at least one year of spontaneous amenorrhea

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal
2. Repeated measurement of supine systolic blood pressure outside the range of 100-140 mm Hg or diastolic blood pressure outside the range of 60-90 mm Hg or pulse less than 55 bpm
3. Any subject with orthostatic hypotension at baseline screening exam
4. Any laboratory value outside the reference range
5. Any evidence of a clinically relevant concomitant disease
6. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic (including insulin-dependent diabetes), immunological or hormonal disorders
7. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders (such as depression) or neurological disorders (such as neuropathy)
8. History of relevant orthostatic hypotension, fainting spells or blackouts
9. Chronic or relevant acute infections
10. History of relevant allergy/hypersensitivity
11. Intake of drugs with a long half-life (greater than 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial.
12. Use of drugs which might reasonably influence the results of the trial within 10 days prior to administration or during the trial
13. Participation in another trial with an investigational drug within two months prior to administration or during the trial
14. Any concomitant therapy
15. Smoker
16. History of alcohol abuse
17. History of drug abuse
18. Blood donation
19. Excessive physical activities (within one week prior to administration or during the trial)
20. Subjects should not swim during the treatment periods of the trial
21. Any condition of the skin, including eczema, psoriasis, or lymphedema, that involves the upper arm in the area that would be utilized for application of the treatments
22. Pregnancy or planning to become pregnant within two months of study completion
23. Positive pregnancy test
24. A screening ECG that displays first-degree atrioventricular block (P-R interval > 0.20 seconds) or other conduction disturbance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 253.2486.1 Boehringer Ingelheim Investigational Site, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in three separate groups.
Groups:
- Catapres®-TTS-3 Crossover 1: TTS-3 Oppanol Then TTS-3 Vistanex: Catapres®-TTS(Transdermal Therapeutic System)-3 (0.3 mg/24 hr) Oppanol® (T1) first, followed by Catapres®-TTS-3 (0.3 mg/24 hr) Vistanex™ (R1). Followed by simultaneous administration of TTS-1 Oppanol® (T2) and TTS-1 Vistanex™ (R2) patches each delivering 0.1mg clinidine/24h.
- Catapres®-TTS-3 Crossover 2: TTS-3 Vistanex Then TTS-3 Oppanol: Catapres®-TTS-3 (0.3 mg/24 hr) Vistanex™ (R1) first, followed by Catapres®-TTS-3 (0.3 mg/24 hr) Oppanol® (T1). Followed by simultaneous administration of TTS-1 Oppanol® (T2) and TTS-1 Vistanex™ (R2) patches each delivering 0.1mg clinidine/24h.
Period: Treatment Period 1(7 Days)
Arm/Group | Catapres®-TTS-3 Crossover 1: TTS-3 Oppanol Then TTS-3 Vistanex | Catapres®-TTS-3 Crossover 2: TTS-3 Vistanex Then TTS-3 Oppanol
Started | 29 | 29
Completed | 28 | 28
Not Completed | 1 | 1
Not completed — Accidental early removal of the patch | 0 | 1
Not completed — Non compliance with the site rule | 1 | 0
Period: Washout Period 1(7 Days)
Arm/Group | Catapres®-TTS-3 Crossover 1: TTS-3 Oppanol Then TTS-3 Vistanex | Catapres®-TTS-3 Crossover 2: TTS-3 Vistanex Then TTS-3 Oppanol
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0
Period: Treatment Period 2 (7 Days)
Arm/Group | Catapres®-TTS-3 Crossover 1: TTS-3 Oppanol Then TTS-3 Vistanex | Catapres®-TTS-3 Crossover 2: TTS-3 Vistanex Then TTS-3 Oppanol
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0
Period: Washout Period 2 (3 Days)
Arm/Group | Catapres®-TTS-3 Crossover 1: TTS-3 Oppanol Then TTS-3 Vistanex | Catapres®-TTS-3 Crossover 2: TTS-3 Vistanex Then TTS-3 Oppanol
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0
Period: Treatment Period 3 (7 Days)
Arm/Group | Catapres®-TTS-3 Crossover 1: TTS-3 Oppanol Then TTS-3 Vistanex | Catapres®-TTS-3 Crossover 2: TTS-3 Vistanex Then TTS-3 Oppanol
Started | 28 | 28
Completed | 28 | 27
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects in the trial were treated and were included in the treated set (TS).
Groups:
- Overall Study: A randomised, double-blind, 2-way crossover design, followed by a period for assessment of adhesive properties of the clonidine patch.
  In the crossover part of the trial, subjects were treated with either Catapres®-TTS delivering 0.3 mg clonidine/24 h (TTS-3) in the Oppanol® formulation (test treatment T1) or Catapres®-TTS-3 (0.3 mg/24 h) with Vistanex™ formulation (reference treatment R1) in each period. In the adhesion phase of the trial, subjects were treated simultaneously with Oppanol® (test treatment T2) and Vistanex™ (reference treatment R2) patches, each delivering 0.1 mg clonidine/24 h (TTS-1).
Arm/Group | Overall Study
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: AUC0-168 (Area Under the Concentration-time Curve of Clonidine in Plasma Over the Time Interval From 0 to 168 h)
Description: AUC0-168 (area under the concentration-time curve of clonidine in plasma over the time interval from 0 to 168 h) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: 1 hour (h) before patch administration and 12h, 24h, 48h, 72h, 96h, 120h, 144h, 168h after patch administration
Population: PKS included all treated subjects who provided at least one observation for at least one primary endpoint without protocol violations with respect to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Groups:
- Catapres®-TTS-3 With Oppanol®: Subject to receive 0.3 mg/24 hr Catapres®-TTS-3 Oppanol® (T1)
- Catapres®-TTS-3 With Vistanex™: Subject to receive 0.3 mg/24 hr Catapres®-TTS-3 Vistanex™ (R1)
Arm/Group | Catapres®-TTS-3 With Oppanol® | Catapres®-TTS-3 With Vistanex™
Number analyzed (Participants) | 52 | 50
pg*h/mL | 82517.99 (19.0) | 80641.47 (19.0)
Statistical Analysis 1: Comparison: Catapres®-TTS-3 With Oppanol® vs Catapres®-TTS-3 With Vistanex™; Test type: Non-Inferiority or Equivalence — The assessment of bioequivalence was based upon 2-sided 90% confidence intervals (CIs) for the ratios of the geometric means Catapres-TTS-3(Oppanol/Vistanex) using an acceptance range of 80.00 to 125.00%; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'Group', 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Mean ratio = 102.33, 90% CI 2-sided [95.74 to 109.37], Standard Error of Mean 19.0 — The estimated value is actually the ratio of Catapres-TTS-3 with Oppanol and Catapres-TTS-3 with Vistanex. The value in parameter dispersion type and dispersion value is actually the intra-individual gCV

2. Primary Outcome: Cavg (Average of Measured Concentrations of Clonidine in Plasma on Days 5, 6, and 7)
Description: Cavg (average of measured concentrations of clonidine in plasma on Days 5, 6, and 7) The values for geometric mean and gCV are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: 1 hour (h) before patch administration and 12h, 24h, 48h, 72h, 96h, 120h, 144h, 168h, 192h, 216h, 240h after patch administration
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Catapres®-TTS-3 With Oppanol® | Catapres®-TTS-3 With Vistanex™
Number analyzed (Participants) | 52 | 50
pg/mL | 697.327 (16.6) | 668.893 (16.6)
Statistical Analysis 1: Comparison: Catapres®-TTS-3 With Oppanol® vs Catapres®-TTS-3 With Vistanex™; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric Means ratio = 104.25, 90% CI 2-sided [98.367 to 110.487], Standard Error of Mean 16.6 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUC0-inf(Area Under the Concentration-time Curve of Clonidine in Plasma Over the Time Interval From 0 to Infinity)
Description: AUC 0-inf(area under the concentration-time curve of clonidine in plasma over the time interval from 0 to infinity) The values for geometric mean and gCV are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Groups:
- Catapres-TTS-3 With Vistanex™: Subject to receive 0.3 mg/24 hr Catapres-TTS-3 Vistanex™ (R1)
Arm/Group | Catapres®-TTS-3 With Oppanol® | Catapres-TTS-3 With Vistanex™
Number analyzed (Participants) | 52 | 50
pg*h/mL | 119127.55 (15.8) | 115903.34 (15.8)
Statistical Analysis 1: Comparison: Catapres®-TTS-3 With Oppanol® vs Catapres-TTS-3 With Vistanex™; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Geometric Means ratio = 102.78, 90% CI 2-sided [97.25 to 108.63], Standard Error of Mean 15.8 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cmax (Maximum Concentration of Clonidine in Plasma)
Description: Cmax (maximum concentration of clonidine in plasma) The values for geometric mean and gCV are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Catapres®-TTS-3 With Oppanol® | Catapres®-TTS-3 With Vistanex™
Number analyzed (Participants) | 52 | 50
pg/mL | 813.516 (16.7) | 781.896 (16.7)
Statistical Analysis 1: Comparison: Catapres®-TTS-3 With Oppanol® vs Catapres®-TTS-3 With Vistanex™; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'Group','sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 104.04, 90% CI 2-sided [98.148 to 110.294], Standard Error of Mean 16.7 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From patch administration until at most 7 days after patch removal, i.e., up to 14 days
Groups:
- TTS-3: Oppanol® (T1): Administration of TTS-3 with Oppanol®
- TTS-3: Vistanex™ (R1): Administration of TTS-3 with Vistanex™
- TTS-1: Vistanex™ (R2) + Oppanol® (T2): Simultaneous administration of TTS-1 with Oppanol® and TTS-1 with Vistanex™
Arm/Group | TTS-3: Oppanol® (T1) | TTS-3: Vistanex™ (R1) | TTS-1: Vistanex™ (R2) + Oppanol® (T2)
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 46/57 | 45/57 | 23/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TTS-3: Oppanol® (T1) (N=57) | TTS-3: Vistanex™ (R1) (N=57) | TTS-1: Vistanex™ (R2) + Oppanol® (T2) (N=56)
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 6 | 4 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 6 | 8 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 1
Application site erythema (General disorders) | 23 | 19 | 10
Application site papules (General disorders) | 12 | 8 | 6
Application site pruritus (General disorders) | 5 | 4 | 0
Fatigue (General disorders) | 3 | 3 | 0
Dizziness (Nervous system disorders) | 4 | 6 | 3
Headache (Nervous system disorders) | 8 | 7 | 3
Insomnia (Psychiatric disorders) | 2 | 4 | 0
Orthostatic hypotension (Vascular disorders) | 11 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.